CLINICAL TRIAL: NCT00174551
Title: The Effect of Prazosin for Nighttime Symptoms of Civilian PTSD
Brief Title: Feasibility Study: The Effect of Prazosin for Nighttime Symptoms of Civilian PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rainier Associates (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20031050
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2005-09

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Prazosin

INTERVENTIONS:
Drug: prazosin

SUMMARY:
Investigating the effect of prazosin for nighttime symptoms of civilian Posttraumatic Stress Disorder.

DETAILED DESCRIPTION:
Each subject will receive prazosin and placebo trials, the order randomized. Day and nighttime symptoms will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* must meet DSM-IV criterion for PTSD

Exclusion Criteria:

* Must not have untreated sleep apnea

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-11; Study Completion 2005-11

PRIMARY OUTCOMES:
Sleep time
REM sleep time
Nightmare frequency
CGI

SECONDARY OUTCOMES:
Distressed Awakenings frequency
PCL-C

CONTACTS AND LOCATIONS:
Overall Officials: Fletcher B Taylor, M.D., Principal Investigator — Rainier Associates
Locations (1):
- Fletcher B. Taylor, Tacoma, Washington, United States